CLINICAL TRIAL: NCT02417129
Title: A Phase III, Randomized, Double-blind, Multi-center, Multi-national Trial to Evaluate Efficacy and Safety of BI 695500 Versus Rituximab as a First-line Immunotherapy Treatment in Patients With Low Tumor Burden Follicular Lymphoma
Brief Title: BI 695500 vs Rituxan First Line Treatment in Patients With Low Tumor Burden Follicular Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1301.6; 2014-004544-36 (EudraCT Number: EudraCT)
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

ARMS (2):
- BI 695500 (Experimental): 375 mg/m2; One intravenous infusion once a week for 4 weeks
  Interventions: Drug: BI 695500
- Rituximab (US reference product) (Active Comparator): 375 mg/m2; One intravenous infusion once a week for 4 weeks
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — BI 695500 375 mg/M2
  Arms: Rituximab (US reference product)
Drug: BI 695500 — BI 695500 375 mg/M2
  Arms: BI 695500

SUMMARY:
This is a Phase III, multicenter, randomized, double-blind, parallel-arm, active comparator trial to evaluate BI 695500 versus rituximab as a first-line immunotherapy treatment in patients with LTBFL. Patients will be randomly assigned in a 1:1 ratio to receive 375 mg/m2 of BI 695500 or rituximab via intravenous (IV) infusion once a week for 4 weeks (total of 4 dosages administered on Days 1, 8, 15, and 22). Disease assessments will be performed at the End of Study (EOS) Visit at Week 30.

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent that is consistent with ICH GCP guidelines and local legislations.
2. Male or female patients, at least 18 years of age at Screening.
3. Histologically-confirmed, stage II - IV NHL (CD20+ FL of Grades 1, 2, or 3a).
4. Low tumor burden according to the GELF criteria
5. Diagnostic biopsies will be centrally reviewed by expert pathologists to confirm correct histology in accordance with WHO guidelines. If the interval since diagnosis is > 12 months, a new biopsy will be required to confirm the histology remained unchanged.
6. Patients not previously treated for their FL, including any previous treatment for FL under clinical trials.
7. ECOG performance status of 0 to 1.
8. Have at least one measurable lesion as per the International Working Group (IWG) criteria 2007 at Screening (lesion clearly measurable in at least two perpendicular dimensions
9. Adequate hematological function (unless abnormalities are related to lymphoma infiltration of the bone marrow) within 28 days prior to randomization
10. Adequate renal and liver function:
11. For participants of reproductive potential (males and females), use of a medically acceptable method of contraception during the trial

Exclusion criteria:

1. Transformation to high-grade lymphoma (secondary to low-grade lymphoma) prior to study entry.
2. Circulating tumor cells = 5 × 109/L.
3. Presence or history of central nervous system lymphoma.
4. Patients receiving current treatment with corticosteroids must not be receiving a dose exceeding 20 mg/day prednisone or equivalent.
5. Patients with prior or concomitant malignancies within 5 years prior to Screening
6. Major surgery within 28 days prior to randomization.
7. Active, chronic or persistent infection that might worsen with immunosuppressive treatment; positive for HIV or tuberculosis (TB) at Screening. Patients who are confirmed positive and those who have active infections are excluded from the trial participation.
8. Patients with serological evidence of HBV infection. Patients seropositive because of HBV vaccine are eligible. HBV positive patients may participate following consultation with a hepatitis expert regarding monitoring and use of HBV antiviral therapy, and provided they agree to receive treatment as indicated.
9. Serious underlying medical conditions, that, per the Investigator¿s discretion, could impair the ability of the patient to participate in the trial.
10. Known hypersensitivity or allergy to murine products.
11. History of a severe allergic reaction or anaphylactic reaction to a biological agent or history of hypersensitivity to any component of the trial medication.
12. Receipt of a live/attenuated vaccine within 12 weeks prior to the Screening Visit.
13. Prior treatment with BI 695500 and/or rituximab.
14. Patients who received any prior therapy using mAbs will be excluded; this does not apply to other biological drugs such as growth factors or anticoagulants.
15. Treatment within a clinical trial within 4 weeks prior to initiation of trial treatment. Patients who have received treatment with a drug that has not received regulatory approval for any indication within 4 weeks or a minimum of 5 half-lives, whichever is longer, of the initial dose of trial medication.
16. Any other co-existing medical or psychological condition(s) that will preclude participation in the trial or compromise ability to give informed consent and/or comply with study procedures.
17. Pregnancy or breast feeding. For women of childbearing potential, a positive serum pregnancy test at the Screening Visit.
18. Patients who have significant cardiac disease, including but not limited to congestive heart failure of Class III or IV of the NYHA classification; uncontrolled angina or arrhythmia; any uncontrolled or severe cardiovascular or cerebrovascular disease; or uncontrolled hypertension.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (21):
- United States (13):
  - Boehringer Ingelheim Investigational Site, Muscle Shoals, Alabama
  - Boehringer Ingelheim Investigational Site, Bakersfield, California
  - Boehringer Ingelheim Investigational Site, Burbank, California
  - Boehringer Ingelheim Investigational Site, Loma Linda, California
  - Boehringer Ingelheim Investigational Site, Albany, Georgia
  - Boehringer Ingelheim Investigational Site, Northbrook, Illinois
  - Boehringer Ingelheim Investigational Site, Pittsfield, Massachusetts
  - Boehringer Ingelheim Investigational Site, Morristown, New Jersey
  - Boehringer Ingelheim Investigational Site, East Setauket, New York
  - Boehringer Ingelheim Investigational Site, Fayetteville, North Carolina
  - Boehringer Ingelheim Investigational Site, Middletown, Ohio
  - Boehringer Ingelheim Investigational Site, Corpus Christi, Texas
  - Boehringer Ingelheim Investigational Site, Ogden, Utah
- Boehringer Ingelheim Investigational Site, Graz, Austria
- Belgium (2):
  - Boehringer Ingelheim Investigational Site, Leuven
  - Boehringer Ingelheim Investigational Site, Namur
- Bulgaria (2):
  - Boehringer Ingelheim Investigational Site, Plovdiv
  - Boehringer Ingelheim Investigational Site, Sofia
- Boehringer Ingelheim Investigational Site, Zagreb, Croatia
- Czechia (2):
  - Boehringer Ingelheim Investigational Site, Brno
  - Boehringer Ingelheim Investigational Site, Prague

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was planned to randomize approximately 250 patients (125 in each treatment group). Actually two patients were randomized, an additional patient was enrolled but not randomized. Two patients were randomised to BI 695500, thus no patient was treated with rituximab in this trial.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that the subject met all strictly implemented inclusion/exclusion criteria.
  Subjects were not to be randomised to trial treatment if any one of the specific entry criteria were violated.
Groups:
- BI 695500: Patients received an infusion of 375 milligram (mg)/square meter (m2) of BI 695500 once a week intravenously for 4 weeks treatment. These 4 dosages were administered on Days 1, 8, 15, and 22 with 26 weeks follow-up.
- Rituximab (US-licensed Rituxan): Patients received an infusion of 375 milligram (mg)/square meter (m2) of rituximab once a week intravenously for 4 weeks treatment. These 4 dosages were administered on Days 1, 8, 15, and 22 with 26 weeks follow-up.
Period: Overall Study
Arm/Group | BI 695500 | Rituximab (US-licensed Rituxan)
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The randomized set (RS) includes all subjects who were randomized to a treatment.
  No patient was randomized to rituximab.
Arm/Group | BI 695500
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.5 (3.54)
Gender [Count of Participants; unit: Participants]
  Female | 2
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Measured as Overall Response Rate (ORR) at Week 30 for BI 695500 Versus Rituximab
Description: The primary objective of this trial was to evaluate statistical equivalence of efficacy as assessed by Overall Response (measured as Overall Response Rate (ORR)) at Week 30 for treatment with BI 695500 versus rituximab (Rituxan®) in patients with untreated low tumor burden follicular lymphoma (LTBFL).
  The overall response measured as Overall Response Rate (ORR), which is the completed response (CR) and the partial response (PR) at Week 30, approximately 26 weeks after the completion of study treatment, as defined by International Working Group (IWG) criteria 2007 via an independent radiology assessment.
  Two patient were randomized and treated with BI 695500, whereas no patient was treated with rituximab in this trial.
Time Frame: From first administration of study medication until 30 weeks thereafter.
Population: As the program was prematurely discontinued and only two patients were randomized at the time of discontinuation, the planned statistical analysis was not performed.
Measure: Number; unit: participants
Arm/Group | BI 695500 | Rituximab (US-licensed Rituxan)
Number analyzed (Participants) | 2 | 0
participants
  CR | 0 |
  PR | 1 |

2. Secondary Outcome: Extrapolated Area Under the Concentration-time Curve of BI 695500 or Rituximab at Steady State Over the Interval 0 Hour (h) to the Next Dose of Trial Medication (AUC0-τ, ss)
Description: Extrapolated area under the concentration-time curve of BI 695500 or rituximab in plasma at steady state over the interval 0 hour (h) to the next dose of trial medication (AUC0-τ, ss) established by population pharmacokinetics.
Time Frame: Sample timepoints Day 1, 8, 22, 23-24 (24-48 hours from start of Cycle 4 infusion), 24-26 (48-96 hours from start of Cycle 4 infusion), 26-36 (96-336 hours from start of Cycle 4 infusion), 78, 134, 204
Population: as for outcome 1
Arm/Group | BI 695500 | Rituximab (US-licensed Rituxan)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Immunogenicity at Week 30
Description: Immunogenicity (rate of anti-drug antibodies) at Week 30 presented as the number of participants having Immunogenicity at Week 30.
  This endpoint was not summarized for arm ' rituximab ', as two patient were randomized and treated with BI 695500, thus no patient was treated with rituximab in this trial.
Time Frame: Day 204 or end of study
Population: Safety Analysis Set (SAF). As the program was prematurely discontinued and only two patients were randomized at the time of discontinuation, the planned statistical analysis was not performed.
Measure: Number; unit: participants
Arm/Group | BI 695500 | Rituximab (US-licensed Rituxan)
Number analyzed (Participants) | 2 | 0
participants | 0 |

ADVERSE EVENTS:
Time Frame: From the first administration of study medication until 26 weeks after the last administration of study medication up to 204 days.
Arm/Group | BI 695500 | Rituximab (US-licensed Rituxan)
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695500 (N=2) | Rituximab (US-licensed Rituxan) (N=0)
Constipation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
Feeling cold (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
As the program was prematurely discontinued and only two patients were randomized at the time of discontinuation, the planned statistical analysis was not performed and safety data are therefore presented in this abbreviated Clinical Trial Report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.